CLINICAL TRIAL: NCT00182546
Title: Canadian Pulmonary Embolism Diagnosis Study
Brief Title: Canadian Pulmonary Embolism Diagnosis Study (CANPEDS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMG-1999-CANPEDS; CIHR-CANPEDS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2005-08

CONDITIONS: Suspected Pulmonary Embolism; Deep Venous Thrombosis
Keywords: Pulmonary Embolism; DVT; Venous Thrombosis; D dimer; DD; Thrombosis; Diagnosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis; Disease

INTERVENTIONS:
Procedure: Two diagnostic management strategies

SUMMARY:
The main objective of the trial is to determine whether D-dimer testing combined with assessment of Pre-Test-Probability (using a standardized clinical model) can be used to markedly simplify the diagnostic process for PE.

It may be safe to omit additional diagnostic testing in selected patients with suspected pulmonary embolism who have a negative D-dimer test

DETAILED DESCRIPTION:
To assess the value of the D-dimer in the diagnosis of PE, we had two sub-groups of patients with suspected PE, low and high pre-test probability. Patients could be randomized either to further or no further testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected PE

Exclusion Criteria:

* Treatment with anticoagulants for greater than 24 hours of performance of D-d
* Comorbid condition limiting survival to less than 3 months
* Absence of acute symptoms within 7 days prior to presentation
* Current pregnancy
* Contraindication to contrast (e.g., allergy, renal failure)
* Geographic inaccessibility which precludes follow-up
* Physician believes patient is inappropriate for study
* failure or inability to provide informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1126
Dates: Start 1998-08; Study Completion 2001-01

PRIMARY OUTCOMES:
DVT or PE during 6 months follow-up

SECONDARY OUTCOMES:
bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MD, PhD, Study Chair — McMaster University; Jeffrey S Ginsberg, MD, Principal Investigator — McMaster University; James Douketis, MD, Principal Investigator — McMaster University; Alexander G Turpie, MB, Principal Investigator — McMaster University; Shannon M Bates, MDCM, Principal Investigator — McMaster University; Mark A Crowther, MD, Principal Investigator — McMaster University; Jeffrey I Weitz, MD, Principal Investigator — McMaster University; Michael Gent, DSc, Principal Investigator — McMaster University; Agnes Y Lee, MD, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - Queen Elizabeth II Health Sciences Ctr., Halifax, Nova Scotia
  - Alexander G. Turpie, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - James Douketis, Hamilton, Ontario
  - HHSC Henderson Campus, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Civic Hospitals, Ottawa, Ontario